CLINICAL TRIAL: NCT00231790
Title: A Multicenter, Double-Blind, Randomized, Placebo-Controlled, Parallel-Group, Dose-Ranging Study of MK0634 in Postmenopausal Women With Overactive Bladder
Brief Title: A Placebo-Controlled Study of MK0634 in Patients With Overactive Bladder (0634-007)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0634-007; 2005_045
Record Dates: First submitted 2005-09-30; First posted 2005-10-04 (Estimated); Last update posted 2015-12-17 (Estimated); Status verified 2015-12

CONDITIONS: Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- MK-0634 50 mg (Experimental): All participants will receive placebo for the 1 week prior to randomization
  Interventions: Drug: MK-0634 50 mg
- MK-0634 125 mg (Experimental): All participants will receive placebo for the 1 week prior to randomization
  Interventions: Drug: MK-0634 125 mg
- MK-0634 375 mg (Experimental): All participants will receive placebo for the 1 week prior to randomization
  Interventions: Drug: MK-0634 125 mg
- Placebo (Placebo Comparator): All participants will receive placebo for the 1 week prior to randomization
  Interventions: Drug: Placebo for MK-0634

INTERVENTIONS:
Drug: MK-0634 50 mg — one capsule orally, once daily in morning
  Other Names: L-000796568
  Arms: MK-0634 50 mg
Drug: MK-0634 125 mg — one or three capsules orally, once daily in morning
  Other Names: L-000796568
  Arms: MK-0634 125 mg; MK-0634 375 mg
Drug: Placebo for MK-0634 — one, two, three or four capsules orally once daily in morning
  Arms: Placebo

SUMMARY:
Overactive bladder is very prevalent in postmenopausal women. The current study is designed to investigate whether a new drug may offer safe and effective treatment.

DETAILED DESCRIPTION:
Clinical development of MK-0634 was discontinued. Study MK-0634-027 was a safety follow-up study to determine if there were any ocular effects of MK-0634 in participants from the United Kingdom who were exposed to MK-0634 during the 007 study.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal females (ages 40-74) with predominantly urge urinary incontinence overactive bladder episodes.
* Patients must meet minimum eligibility requirements (e.g., average number of micturitions/day) based on screening diary cards.

Exclusion Criteria:

* Patients must not suffer from diabetes insipidus
* Hyperglycemia
* Hypercalcemia
* Orthostatic hypotension
* Active/recurrent urinary tract infections (>6 episodes per year)
* Patients must be willing to discontinue their current OAB medication therapy.

Ages: 40 Years to 74 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 848 (Actual)
Dates: Start 2005-08; Primary Completion 2006-09 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the number of micturitions per day averaged over a diary card week (4 to 10 days) | Baseline and Week 8
Proportion of participants with abnormal retinal photography (Follow-up Study 007 only) | Day 1 of Follow-up
Proportion of participants with abnormal visual field test (Follow-up Study 007 only) | Day 1 of Follow-up

SECONDARY OUTCOMES:
Change from baseline in the number of total incontinence episodes | Baseline and Week 8
Number of urge-incontinence episodes | Up to 8 weeks
Number of urgency episodes per day averaged over a diary card week (4 to 10 days) | up to 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC